CLINICAL TRIAL: NCT00243061
Title: A Phase II Study of AZD2171 in Previously Untreated Patients With Metastatic or Recurrent Malignant Melanoma
Brief Title: AZD2171 in Treating Patients With Recurrent or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03026; PHL-038 (Other Grant/Funding Number: N01CM62203); N01CM62203 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Acral Lentiginous Malignant Melanoma; Ciliary Body and Choroid Melanoma, Medium/Large Size; Ciliary Body and Choroid Melanoma, Small Size; Extraocular Extension Melanoma; Intraocular Melanoma; Iris Melanoma; Lentigo Maligna Malignant Melanoma; Recurrent Melanoma; Stage, Intraocular Melanoma; Stage IV Melanoma; Superficial Spreading Malignant Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with recurrent or stage IV melanoma. AZD2171 may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective tumor response rate of AZD2171 administered to patients with recurrent or metastatic malignant melanoma.

II. To assess the toxicity, median survival time, 1-year survival rate, response or stable disease duration, time to disease progression and clinical benefit response of AZD2171 administered to patients with recurrent or metastatic malignant melanoma.

III. To measure baseline and post-treatment levels of angiogenic growth factors and receptors, as well as circulating endothelial cells, and to explore the relationship between these potential correlative endpoints and clinical outcome.

IV. To assess changes in blood flow and vessel permeability using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) pre- and post-treatment, and to explore the relationship between these potential imaging endpoints and clinical outcome.

V. To look for polymorphisms of kdr/flk-1, and other genes in this pathway, by performing pharmacogenetic analysis of pbmc's, and correlate genotype with VEGF levels and response to therapy.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed recurrent/metastatic malignant melanoma (stage IV acral lentiginous, lentigo maligna, superficial spreading or ocular malignant melanoma)
* Measurable disease- at least 1 lesion accurately measured in at least 1 dimension (longest diameter) as >=20mm with conventional techniques or >=10mm with spiral CT scan

  * Previously irradiated lesions not considered measurable unless they demonstrated progression prior to study entry
* No prior chemotherapy (including regional therapy); prior adjuvant immunotherapy permitted if completed >3 months prior to study entry; patients may have received prior radiation therapy if completed >=4 weeks prior to study entry

  * Previous surgery permissible if performed >=4 weeks prior to study entry
* Life expectancy >12 weeks
* ECOG performance status=< 2 (Karnofsky>=60%)
* Leukocytes>=3,000/mcL
* Absolute neutrophil count>=1,500/mcL
* Platelets>=100,000/mcL
* Hemoglobin>=8g/dL
* Total bilirubin<1.5x institutional ULN (IULN)
* AST/ALT=<3 x IULN (5xULN if liver metastases)
* Creatinine within IULN
* Creatinine within IULN OR
* Creatinine clearance>=60mL/min/m^2 if creatinine levels above IULN
* Baseline blood pressure <140/90mmHg; may be taking antihypertensive medications
* AZD2171 has shown to terminate fetal development in rat as expected for process dependent on VEGF signaling; women of childbearing potential must have negative pregnancy test prior to study entry; women of childbearing potential/men must agree to use adequate contraception (hormonal/barrier method of birth control; abstinence) prior to study entry and for duration of study
* Ability to understand/willingness to sign written informed consent

Exclusion Criteria:

* Any previous chemotherapy or immunotherapy for recurrent/metastatic disease; patients who have had radiotherapy or major surgery within 4 weeks prior to entering study or those who have not recovered from AEs due to treatment received more than 4 weeks earlier
* May not be concurrently receiving other investigational agents nor have participated in an investigational trial of bio-, chemo- or immunotherapy agents
* Known brain metastases because of their poor prognosis and because patients often develop progressive neurologic dysfunction that would confound evaluation of neurologic and other AEs
* History of allergic reactions attributed to compounds of similar chemical/biologic composition to AZD2171
* Mean QTc>470msec (Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome
* >+1 proteinuria on 2 consecutive dipsticks taken no less than 1 week apart
* Uncontrolled intercurrent illness including but not limited to hypertension, ongoing/active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women excluded from study because AZD2171 is a VEGF inhibitor with known abortifacient effects; breastfeeding should be discontinued if mother is treated with AZD2171
* HIV-positive patients on combination antiretroviral therapy are ineligible because of potential for PK interactions with AZD2171; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Any significant abnormality noted in ECG within 14 days of treatment
* A NYHA classification of III or IV (NOTE: Patients classified as class II controlled with treatment may continue with increase monitoring)
* Conditions requiring concurrent use of drugs/biologics with proarrhythmic potential; these drugs are prohibited during studies with AZD2171

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine McWhirter, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cediranib Maleate): Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cediranib maleate: Given orally
  laboratory biomarker analysis: Correlative studies
  dynamic contrast-enhanced magnetic resonance imaging: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 67 [28 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Region of Enrollment [Number; unit: participants]
  Canada | 10
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response (Partial or Complete Response) According to RECIST
Description: Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [J Nat Cancer Inst 92(3):205-216, 2000]. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions, assessed by CT or MRI; Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: Up to 6 years
Population: Out of 24 patients analyzed, 0 patients had objective response of PR or CR as defined by RECIST
Measure: Number; unit: participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 24
participants | 0

2. Primary Outcome: Prolonged Stable Disease According to RECIST
Time Frame: Up to 6 months
Measure: Number; unit: participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 24
participants | 9

3. Secondary Outcome: Median Survival Time
Time Frame: Up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 24
months | 9.9 [6.8 to 20.6]

4. Secondary Outcome: Survival Rate
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 24
percentage of participants | 41 [24 to 64]

5. Secondary Outcome: Response Duration
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 6 years
Population: None of the patients had Partial or complete response
Measure: Number; unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 24
months | 0

6. Secondary Outcome: Stable Disease Duration
Time Frame: From the start of the treatment until the criteria for progression are met, assessed up to 6 years
Population: Only 17 of the 24 accrued patients were evaluable for response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 17
months | 4.6 [3.1 to 9.1]

7. Secondary Outcome: Highest Toxicity Grade Assessed by NCI CTCAE Version 3.0
Time Frame: Up to 6 years after completion of treatment
Measure: Number; unit: highest grade
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 23
highest grade | 4

8. Secondary Outcome: Time to Disease Progression
Time Frame: Up to 6 years
Population: 9 patients developed progressive disease
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 24
months | 4.1 [1.8 to 7.4]

9. Secondary Outcome: Clinical Benefit Response
Time Frame: Up to 6 years
Population: data were not collected
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

10. Secondary Outcome: Changes in Levels of Soluble Angiogenic Factors
Time Frame: From baseline to up to 6 years
Population: data were not collected
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Vessel Permeability and Blood Flow by DCE-MRI
Time Frame: From baseline to up to 28 days after starting daily oral dosing
Population: data were not collected
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Cediranib Maleate)
Serious Adverse Events (participants affected / at risk) | 9/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cediranib Maleate) (N=24)
Hypertension (Vascular disorders) | 3
Non-cardiac chest pain (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Dysphasia (Nervous system disorders) | 1
Blurred vision (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cediranib Maleate) (N=24)
Fatigue (General disorders) | 19
Diarrhea (Gastrointestinal disorders) | 18
Hypertension (Vascular disorders) | 17
Hyperglycemia (Metabolism and nutrition disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less